CLINICAL TRIAL: NCT04364594
Title: Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2): Diagnostic Targets for Customized Medicine.
Brief Title: COVID-19 Search in Conjunctival Cells
Acronym: COVID-T
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0013008/20
Record Dates: First submitted 2020-04-22; First posted 2020-04-28 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: COVID 19; Pulmonary Disease
Keywords: Conjunctival swabs; Diagnosis; SARS-CoV2; Systemic Impairment
MeSH Terms: conditions — COVID-19; Lung Diseases; Disease | interventions — Radiation; Tomography, X-Ray Computed; Radionuclide Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- affected individual (Experimental): Patients affected by Coronavirus 19 admitted to the hospital setting
  Interventions: Diagnostic Test: conjunctival swab

INTERVENTIONS:
Diagnostic Test: conjunctival swab — analysis of conjunctival cells (real time PCR) collected by conjunctival swabs in both eyes
  Other Names: Pulmonary involvement determined by X-Ray (XR) rays and Computed Tomography (CT) scan

SUMMARY:
The patients enrolled in this study will be all patients entering triage with suspicion of SARS-CoV2. Planned activities are required by the nasopharyngeal swab in parallel with the analysis of the conjunctival swab to identify new potential alternative and equally effective diagnostic pathways.

Simultaneously systemic data (as Pulmonary images, hematological parameters etc.) will be collected to observe a possible correlation between conjunctival swab positivity and systemic impairment.

DETAILED DESCRIPTION:
In recent months, considerable interest has turned to Coronavirus infection in terms of early diagnosis and targeted therapy. Thanks to the experimentation of new therapeutic strategies, it becomes more and more evident how some subgroups of patients can benefit from a specific treatment, while others would have no benefit.

Alongside these innovative clinical research techniques, early diagnosis that would lead to identifying those at risk of a new disease and new infection is becoming increasingly important.

COVID-19 occurred in China in December 2019 but probably already had an expression in the previous months. The number of victims reached its peak in January 2020 with prevalent involvement of patients already at risk or with previous physical debilitations. But even apparently healthy and young individuals can be affected by infections with a lethal outcome. Since January 2020 new cases have been registered all over the world and prevalently in Italy. The main way of infection identified is the respiratory tract, but infection through conjunctival may not be excluded.

The main outcome of this research is to investigate the positivity of the COVID-19 virus in the conjunctival mucosa to establish a new diagnostic target.

All patients will receive both the conjunctival swab and nasopharyngeal swab. The conjunctival swab will be performed in each eye and both swabs will be inserted into the same virus test tube. The swab samples will be sent in the same day to the microbiology laboratory for examination by Real Time-PCR.

The secondary outcome will be to evaluate the possible positivity of the conjunctival swab with the degree of systemic impairment. This objective has the purpose of personalized medicine.

ELIGIBILITY:
Inclusion Criteria:

* All patients accepted to triage with positivity or suspected positivity to COVID-19 will be enrolled in the study and both conjunctival and nasopharyngeal swab will be performed.

Exclusion Criteria:

* To date, there are no exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-03-26 (Actual); Primary Completion 2020-04-24 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
Conjunctival swab results based on RT-PCR | 2 months
  Collection of conjunctival cell samples from eyes of COVID-19 patients. Analysis of conjunctival cells by real-time PCR to document presence of COVID-19. Binary outcome: yes, no. To evaluate the result in relation to nasopharyngeal swab (binary outcome yes, no) and to correlate conjunctival with nasopharyngeal swab positivity

SECONDARY OUTCOMES:
Conjunctival swab positivity in relation to Pulmonary and blood abnormalities | 2 months
  To evaluate the agreement between conjunctival swab positivity and the degree of systemic impairment. The latter will be measured on the basis of pulmonary disease severity as assessed by a standardized scale (Occhipinti et al 2019) for interstitial lung involvement in systemic sclerosis; the blood measurements of d-dimer, LDH and reactive CP.

CONTACTS AND LOCATIONS:
Locations (1):
- Maria Cristina Savastano, Roma, Italy

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol approved by Ethical Committee, informed consent, clinical study report, will be available
Supporting Information: Study Protocol, ICF, CSR
Time Frame: The data will be available immediately after the statistical analysis of the results and will remain available for at least 1 year
Access Criteria: On request by e-mail

REFERENCES:
- [Background] Occhipinti M, Bosello S, Sisti LG, Cicchetti G, de Waure C, Pirronti T, Ferraccioli G, Gremese E, Larici AR. Quantitative and semi-quantitative computed tomography analysis of interstitial lung disease associated with systemic sclerosis: A longitudinal evaluation of pulmonary parenchyma and vessels. PLoS One. 2019 Mar 12;14(3):e0213444. doi: 10.1371/journal.pone.0213444. eCollection 2019. PMID 30861018